CLINICAL TRIAL: NCT00687388
Title: The Clinical Efficacy of Non-steroidal Anti-inflammation Drugs in Patients With Benign Prostatic Hyperplasia: A Prospective Randomized Multicenter Trial
Brief Title: The Clinical Efficacy of Non-steroidal Anti-inflammation Drugs in Patients With Benign Prostatic Hyperplasia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: in order to prepare a new clinical trial to evaluate with pathological change
Sponsor: Samsung Medical Center (Other)
Collaborators: The Korean Urological Association (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-07-084
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Cyclooxygenase 2 Inhibitors; Alpha Blockers; Treatment Outcome
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; alfuzosin; Doxazosin; Terazosin; Celecoxib; Adrenergic alpha-Antagonists; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alpha-blocker (Active Comparator): Alpha-blocker only
  Interventions: Drug: selective alpha 1-blockers
- NSAID (Active Comparator): NSAID only
  Interventions: Drug: celecoxib
- alpha-blocker and NSAID (Experimental): Combination treatment of alpha-blocker and NSAID
  Interventions: Drug: alpha-blocker and NSAID

INTERVENTIONS:
Drug: selective alpha 1-blockers — Continued medication that the patient had before the enrollment of this study (tamsulosin 0.2mg, alfuzosin 10mg, doxazosin 4, 8mg, or terazosin 2-10mg daily for 8 weeks)
  Other Names: tamsulosin; alfuzosin; doxazosin; terazosin
  Arms: Alpha-blocker
Drug: celecoxib — 200mg daily for 8 weeks
  Arms: NSAID
Drug: alpha-blocker and NSAID — amsulosin 0.2mg, alfuzosin 10mg, doxazosin 4, 8mg, or terazosin 2-10mg daily for 8 weeks and celecoxib 200mg daily for 8 weeks
  Other Names: tamsulosin and celecoxib; alfuzosin and celecoxib; doxazosin and celecoxib; terazosin and celecoxib
  Arms: alpha-blocker and NSAID

SUMMARY:
Non-steroidal Anti-inflammation Drugs can effectively reduce the lower urinary tract symptoms from benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Who had the treatment of BPH with alpha-1 blockers for more than 3 months
* Who have the IPSS(International Prostatic Symptom Score) >= 15
* Who have the maximum flow rate(Qmax) < 15 with voided volume > 150mL
* Who have the PPBC(patient's perception of bladder condition) >= 3 (The PPBC was assessed by the use of a six point ordered categorical scale(1-6 point). The higher score means the higher bother)
* Who had the PSA level < 4 ng/mL within 6 months (But, the patient who are revealed not to have prostate cancer by prostate biopsy can be included even if he had PSA level of 4-10 ng/mL)
* Who underwent the transrectal ultrasound of prostate within 6 months
* Who can understand this study and can give the informed consent

Exclusion Criteria:

* Who had regular intake of 5-alpha reductase inhibitor or NSAID within 6 months before screening
* Who have peptic ulcer and/or asthma
* Who have urologic malignancies such as prostate cancer and bladder cancer
* Who have urethral strictures, large bladder diverticuli, and bladder neck contractures
* Who had surgical treatment for BPH
* Who have histories of bladder and/or urethra
* Who have serum PSA level more than 10 ng/ml
* Who have histories of orthostatic hypotension
* Who have serum creatinine level more than 2.0 mg/dl
* Who have serum ALT and/or AST level more than 1.5 times of normal upper limit
* Who have heart failure
* Who have histories of bacterial prostatitis within 1 year
* Who have histories of active urinary tract infection within 1 month
* Who have histories of the biopsy of bladder and prostate within 1 month
* Who are unable to void
* Who use pads because of incontinences
* Who have hypersensitivities for alpha blockers that include quinazoline, NSAID, aspirin, sulfonamide
* Who have histories of unstable angina, myocardial infarction, and cerebrovascular accident within 6 months
* Who have neurogenic bladder due to multiple sclerosis, Parkinson's disease, Spinal injuries and etc.
* Who have thinking disturbances
* Who have histories of abuses of alcohol and/or other drugs
* Who seem to be not fit to this study by the decision of investigators

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The changes of International Prostatic Symptom Scores after medications | 8 weeks

SECONDARY OUTCOMES:
The changes of voiding frequencies after medications | 8 weeks
The changes of 'ICS male questionnaire-short form' after medications | 8 weeks
Patient perception of treatment benefit questionnaire | 8 weeks
The changes of 'patient perception of bladder condition' after medications | 8 weeks
The changes of maximum flow rate and postvoid residuals after medications | 8 weeks
The changes of serum PSA levels after medications | 8 weeks
The changes of WBC counts on the expressed prostatic secretions after medications | 8 weeks
Complications | During all study periods

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D., M.D., Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Background] Kramer G, Steiner GE, Handisurya A, Stix U, Haitel A, Knerer B, Gessl A, Lee C, Marberger M. Increased expression of lymphocyte-derived cytokines in benign hyperplastic prostate tissue, identification of the producing cell types, and effect of differentially expressed cytokines on stromal cell proliferation. Prostate. 2002 Jun 1;52(1):43-58. doi: 10.1002/pros.10084. PMID 11992619
- [Background] Untergasser G, Madersbacher S, Berger P. Benign prostatic hyperplasia: age-related tissue-remodeling. Exp Gerontol. 2005 Mar;40(3):121-8. doi: 10.1016/j.exger.2004.12.008. Epub 2005 Jan 22. PMID 15763388
- [Background] Lee KL, Peehl DM. Molecular and cellular pathogenesis of benign prostatic hyperplasia. J Urol. 2004 Nov;172(5 Pt 1):1784-91. doi: 10.1097/01.ju.0000133655.71782.14. PMID 15540721
- [Background] Handisurya A, Steiner GE, Stix U, Ecker RC, Pfaffeneder-Mantai S, Langer D, Kramer G, Memaran-Dadgar N, Marberger M. Differential expression of interleukin-15, a pro-inflammatory cytokine and T-cell growth factor, and its receptor in human prostate. Prostate. 2001 Dec 1;49(4):251-62. doi: 10.1002/pros.10020. PMID 11746271
- [Background] Kakehi Y, Segawa T, Wu XX, Kulkarni P, Dhir R, Getzenberg RH. Down-regulation of macrophage inhibitory cytokine-1/prostate derived factor in benign prostatic hyperplasia. Prostate. 2004 Jun 1;59(4):351-6. doi: 10.1002/pros.10365. PMID 15065082
- [Background] Steiner GE, Newman ME, Paikl D, Stix U, Memaran-Dagda N, Lee C, Marberger MJ. Expression and function of pro-inflammatory interleukin IL-17 and IL-17 receptor in normal, benign hyperplastic, and malignant prostate. Prostate. 2003 Aug 1;56(3):171-82. doi: 10.1002/pros.10238. PMID 12772186
- [Background] Wang W, Bergh A, Damber JE. Chronic inflammation in benign prostate hyperplasia is associated with focal upregulation of cyclooxygenase-2, Bcl-2, and cell proliferation in the glandular epithelium. Prostate. 2004 Sep 15;61(1):60-72. doi: 10.1002/pros.20061. PMID 15287094
- [Background] Kramer G, Marberger M. Could inflammation be a key component in the progression of benign prostatic hyperplasia? Curr Opin Urol. 2006 Jan;16(1):25-9. PMID 16385197
- [Background] Rohrmann S, De Marzo AM, Smit E, Giovannucci E, Platz EA. Serum C-reactive protein concentration and lower urinary tract symptoms in older men in the Third National Health and Nutrition Examination Survey (NHANES III). Prostate. 2005 Jan 1;62(1):27-33. doi: 10.1002/pros.20110. PMID 15389816
- [Background] Araki T, Yokoyama T, Kumon H. Effectiveness of a nonsteroidal anti-inflammatory drug for nocturia on patients with benign prostatic hyperplasia: a prospective non-randomized study of loxoprofen sodium 60 mg once daily before sleeping. Acta Med Okayama. 2004 Feb;58(1):45-9. doi: 10.18926/AMO/32115. PMID 15157011